CLINICAL TRIAL: NCT02903446
Title: Denosumab In Addition To Intense Urate-Lowering Therapy for Bone Erosions in Gout: A Pilot Study
Brief Title: Denosumab In Addition To Intense Urate-Lowering Therapy for Bone Erosions
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: University of Auckland, New Zealand (Other)
Responsible Party: Principal Investigator, Angelo L. Gaffo, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F160315004
Record Dates: First submitted 2016-09-13; First posted 2016-09-16 (Estimated); Results first posted 2021-08-31 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): Denosumab 60 mg administered subcutaneously (SC) every 6 months for a year + urate lowering therapy (ULT) standard of care
  Interventions: Drug: Denosumab
- Control (No Intervention): Standard urate lowering therapy

INTERVENTIONS:
Drug: Denosumab — Participants will be randomized (1:1) allocation to denosumab 60 mg administered subcutaneously (SC) every 6 months for a year + ULT standard of care OR ULT standard of care therapy
  Other Names: Prolia
  Arms: Intervention

SUMMARY:
Bone erosions are a common manifestation and feature of structural damage in severe/chronic tophaceous gout. Management of this destructive and often debilitating gout complication has focused exclusively on urate-lowering therapy (ULT) to reduce frequency of gout attacks, but little attention has been given to prevention or reversal of gout related bone erosions and other structural damage to bone caused by gout. Since there is no known effective treatment to attenuate or improve structural damage caused by gout, we propose a pilot, controlled, proof-of-concept study in which denosumab, an FDA approved medication for the treatment of bone loss, will be added to standard ULT in 20 patients with erosive gout.

DETAILED DESCRIPTION:
A recently published clinical trial with zoledronic acid failed to show an effect in improving bone erosions among individuals with chronic tophaceous gout, despite improvements in bone mineral density (BMD) and bone turnover markers. However, it is known that increased numbers of osteoclasts (cells that absorb bone tissue during growth and healing) in patients with tophaceous gout are most likely a result of enhanced osteoclast activity as these patients also have higher circulating levels of the protein receptor activator of nuclear factor kappa-B ligand (RANKL). RANKL has been identified to affect the immune system and control bone regeneration and remodeling.

Furthermore, peripheral blood cells and synovial fluid cells taken from patients with erosive gout preferentially formed osteoclast-like cells in the presence of RANKL. The number of osteoclasts formed significantly correlates with the number of tophi in gout patients.

Denosumab (Prolia®) is a fully human monoclonal antibody with a high affinity for RANKL that can bind and neutralize the activity of human RANKL. Given the relevance of RANKL in the mechanism of gouty erosions,a central hypothesis of this pilot study is that denosumab is more likely to precisely target RANKL and the mechanism of gouty erosions than zoledronic acid.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 years or older and able to provide informed consent
* Diagnosis of gout according to the American College of Rheumatology (ACR) / European League Against Rheumatism (EULAR) classification criteria
* Radiographic foot bone erosion attributable to gout and confirmed by a radiologist
* Serum urate of ≤ 5 mg/dL (300 µmol/L) or less*

Exclusion Criteria:

* Treatment with bisphosphonates in the preceding 2 years
* Any prior treatment with denosumab
* Women of childbearing potential, who are not currently using birth control, are pregnant, planning to become pregnant, or are breast-feeding
* Men planning to conceive in the next 12 months
* Unstable systemic medical condition
* Uncontrolled hyperthyroidism
* Uncontrolled hypothyroidism
* History of Addison disease
* History of osteomalacia
* History of osteonecrosis of the jaw (ONJ)
* History of atypical femur fracture
* History of tooth extraction, jaw surgery, dental implants, or other dental surgery within the prior 6 months
* History of anorexia nervosa, bulimia (by history or physical) or obvious malnutrition.
* Invasive dental work planned in the next 2 years
* History of Paget's disease of bone
* Other bone diseases which affect bone metabolism
* Vitamin D deficiency [25(OH) vitamin D level < 20 ng/mL (<49.9 nmol/L)]†
* Hypercalcemia
* Elevated transaminases ≥ 2.0 x upper limit of normal (ULN)
* Elevated total bilirubin > 1.5x ULN
* History of any solid organ or bone marrow transplant
* Malignancy within the last 5 years (except cervical carcinoma in situ or basal cell carcinoma)
* Hypocalcemia
* Poorly tolerant of ULT including allopurinol, febuxostat, or probenecid
* Estimated glomerular filtration rate < 30 mL/minute/1.73 m^2
* Current use of any biological therapy (eg. infliximab, etanercept, adalimumab, etc.)
* Treatment history with pegloticase or another recombinant uricase
* Recipient of an investigational drug within 4 weeks prior to study drug administration or plans to take an investigational agent during the study

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential study participants were screened for enrollment at rheumatology clinics located at the University of Alabama at Birmingham and the University of Auckland. Participants were recruited between March 2017 and May 2019.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (15) | 63 (9.4) | 65.0 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 9 | 10 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  European descent | 6 | 5 | 11
  Maori | 0 | 2 | 2
  Asian | 1 | 1 | 2
  Pacific Islander | 0 | 0 | 0
  Other | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 4 | 9
  New Zealand | 5 | 6 | 11
Serum Urate [Mean (Standard Deviation); unit: mg/dL] | 4.3 (0.5) | 4.2 (0.7) | 4.3 (0.6)
Estimated glomerular filtration rate [Mean (Standard Deviation); unit: mL/min/1.73m2] | 76.5 (32) | 72 (15.3) | 74.2 (24.5)
CT Erosion Score (range 0-140 total of 14 bones) [Mean (Standard Deviation); unit: units on a scale] — Change in the foot CT bone erosion score from baseline to 12 months. A total of 14 bones of the foot are scored. Each bone of the scored separately on a scale from 0 to 10, based on the proportion of eroded bone compared with the 'assessed bone volume', judged on all available images-0: no erosion; 1: 1-10% of bone eroded; 2: 11-20%, etc.
  Higher score indicate worsening of erosion.
  units on a scale | 6.6 (5.4) | 7.0 (5.1) | 6.8 (5.1)
Serum CTX [Mean (Standard Deviation); unit: pg/mL] — Measure of the amount carboxy-terminal collagen crosslinks (CTX) in serum
  pg/mL | 316.6 (152.6) | 286.9 (111.5) | 303.4 (133.0)
Health Assessment Questionnaire -Disability Index Total (range from 0-3.0) [Mean (Standard Deviation); unit: HAQ Score] — 0 to 1 are generally considered to represent mild to moderate difficulty, 1 to 2 moderate to severe disability, and 2 to 3 severe to very severe disability.
  HAQ Score | 0.36 (0.61) | 0.39 (0.44) | 0.38 (0.52)
Short Form Survey (SF-12) physical component score (range 0-100) [Mean (Standard Deviation); unit: SF-12 score] — The SF-12 measures eight concepts commonly represented in widely used surveys: physical functioning. Subject reported change in physical and mental health by Short Form Health Survey (SF-12) scores assessed from baseline over 12 months. Range 0-100 with higher scores representing better self-reported health.
  SF-12 score | 43.6 (11.9) | 43.9 (7.3) | 43.8 (9.6)
Short Form Survey (SF-12) mental component score (range 0-100) [Mean (Standard Deviation); unit: SF-12 score] — Subject reported change in physical and mental health by Short Form Health Survey (SF-12) scores assessed from baseline over 12 months. Range 0-100 with higher scores representing better self-reported health.
  SF-12 score | 57.5 (4.2) | 55.1 (10.4) | 56.3 (7.8)
Visual Analogue Pain Score (range 0-10) [Mean (Standard Deviation); unit: visual analog pain scale] — A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values (0-10)
  visual analog pain scale | 2.2 (3.7) | 1.3 (1.5) | 1.8 (2.9)

OUTCOME MEASURES:

1. Primary Outcome: CT Bone Erosion Score
Description: Change in the foot CT bone erosion score from baseline to 12 months. A total of 14 bones of the foot are scored. Each bone of the scored separately on a scale from 0 to 10, based on the proportion of eroded bone compared with the 'assessed bone volume', judged on all available images-0: no erosion; 1: 1-10% of bone eroded; 2: 11-20% bone eroded; 3:21-30% of bone eroded; 4: 31-40% of bone eroded; 5: 51-60% bone eroded; 7:61-70% of bone eroded; 8: 71-80% of bone eroded; 9: 81-90% bone eroded; 10:>=91% of bone eroded.
  Higher score indicates worsening of erosion. Score ranges from 0 to 140.
Time Frame: Baseline, 12 months
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 10 | 10
Score on a scale | 6.6 (5.4) | 7.0 (5.1)

2. Secondary Outcome: Decrease in Bone Reabsorption
Description: Change in bone reabsorption as measured by serum carboxy-terminal collagen crosslinks (CTX) levels (pg/mL) over 12 months. Lower values represent varying degrees of suppression of normal bone turnover.
  The reference ranges for C-terminal telopeptide in serum are as follows:
  Female (premenopausal): 40-465 pg/mL Female (postmenopausal): 104-1008 pg/mL Male: 60-700 pg/mL
Time Frame: Baseline, 12 months
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Intervention | Control
Number analyzed (Participants) | 10 | 10
pg/mL | 177.6 (143.1) | 324.1 (113.3)

3. Secondary Outcome: Change in Subject Reported Functional Status (Disability)
Description: Change in subject reported functional status (disability) by Health Assessment Questionnaire (HAQ) will be assessed from baseline over 12 months. 0 to 1 are generally considered to represent mild to moderate difficulty, 1 to 2 moderate to severe disability, and 2 to 3 severe to very severe disability.
Time Frame: Baseline, 12 months
Measure: Mean (Standard Deviation); unit: Difference in HAQ score from baseline
Arm/Group | Intervention | Control
Number analyzed (Participants) | 10 | 10
Difference in HAQ score from baseline | .33 (.30) | .11 (0.24)

4. Secondary Outcome: Subject Reported Change in Physical Health
Description: Subject reported change in physical and mental health by Short Form Health Survey (SF-12) scores assessed from baseline over 12 months. Range 0-100 with higher scores representing better self-reported health.
Time Frame: Baseline, 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 10 | 10
units on a scale | 45.5 (12.6) | 52.3 (1.8)

5. Secondary Outcome: Subject Reported Change in Mental Health
Description: Subject Reported Change in Mental Health on SF-12 mental component form. Range 0-100 with higher scores representing better self-reported health
Time Frame: Baseline, 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 10 | 10
units on a scale | 58.7 (6.7) | 53.1 (7.6)

6. Secondary Outcome: Assessment of Pain
Description: Assessment of pain score by visual analogue scale (VAS) reported from baseline over 12 months. Range 0-10 with higher scores representing more pain.
Time Frame: Baseline, 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 10 | 10
units on a scale | 1.3 (3.1) | 1.2 (1.4)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 5/10 | 6/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=10) | Control (N=10)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Gastro-esophageal reflux (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomitting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophageal refulx (Gastrointestinal disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Skin Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-26): https://cdn.clinicaltrials.gov/large-docs/46/NCT02903446/Prot_SAP_000.pdf